CLINICAL TRIAL: NCT07327788
Title: Iparomlimab and Tuvonralimab (QL1706) With Bevacizumab and RALOX Hepatic Arterial Infusion Chemotherapy for Hepatocellular Carcinoma (HCC) With Vp3/4 Portain Vein Thrombosis : A Prospective, Multicenter, Phase II Study
Brief Title: QL1706 in Combination With Bevacizumab and RALOX HAIC for Hepatocellular Carcinoma With Vp3/4 PVTT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2025-646
Record Dates: First submitted 2025-12-25; First posted 2026-01-08 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Hepatecellular Carcinoma; RALOX-HAIC（Hepatic Arterial Infusion Chemotherapy With Raltitrexed and Oxaliplatin; Bevacizumab; Type VP3/4 Portal Vein Tumor Thrombosis; Iparomlimab and Tuvonralimab Injection; QL1706
MeSH Terms: interventions — Bevacizumab; raltitrexed; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Iparomlimab and Tuvonralimab Injection (QL1706) combined with Bevacizumab plus RALOX-HAIC (Experimental)
  Interventions: Drug: Iparomlimab and Tuvonralimab Injection (QL1706); Drug: Bevacizumab; Procedure: Hepatic Arterial Infusion Chemotherapy with Raltitrexed and Oxaliplatin (RALOX-HAIC)

INTERVENTIONS:
Drug: Iparomlimab and Tuvonralimab Injection (QL1706) — Iparomlimab and Tuvonralimab Injection (QL1706)will be administered at a dose of 7.5 mg/kg via intravenous infusion (no premedication required). Each infusion shall last for 30 minutes (no less than 20 minutes and no more than 60 minutes), with an administration interval of 3 weeks, and one treatment cycle is defined as 3 weeks. The maximum cumulative treatment duration shall be 2 years. The administration window for QL1706 is within 7 days after hepatic arterial infusion chemotherapy. If the administration is delayed beyond the scheduled time, the dose for this cycle will be omitted, and the subsequent administration will be resumed at the original dose in accordance with the next scheduled time.
Drug: Bevacizumab — Bevacizumab will be administered at a dose of 15 mg/kg via intravenous infusion (no premedication required), once every 3 weeks, with one treatment cycle defined as 3 weeks. The maximum cumulative treatment duration shall be 2 years.
Procedure: Hepatic Arterial Infusion Chemotherapy with Raltitrexed and Oxaliplatin (RALOX-HAIC) — RALOX regimen chemotherapy will be delivered via hepatic arterial infusion (HAIC). The procedure will be performed using the Seldinger technique for femoral artery puncture and catheterization. Digital subtraction angiography (DSA) will be conducted to identify the blood supply artery of the lesion. A conventional catheter (or a microcatheter if necessary) will be superselectively inserted into the tumor-feeding artery via the celiac trunk or superior mesenteric artery, then the catheter will be retained in the catheter sheath and fixed to the body surface before the patient is returned to the ward. In the ward, the catheter will be connected to an infusion pump for continuous infusion of the following chemotherapeutic agents: Oxaliplatin 85 mg/m² over 2 to 4 hours, and Raltitrexed 3 mg/m² over 1 to 2 hours. The catheter will be removed upon completion of chemotherapy, followed by compression bandaging for hemostasis for 6 hours.

SUMMARY:
The goal of this prospective, single-arm, multi-center Phase II clinical trial is to evaluate the clinical efficacy and safety of QL1706 combined with bevacizumab and RALOX hepatic artery infusion chemotherapy in treating liver cancer patients with VP3/4 portal vein tumor thrombus. It will also explore molecular biomarkers that predict the efficacy of this combined therapy.

The main questions it aims to answer are:

What is the progression-free survival (PFS) of patients treated with this regimen? What are the objective response rate (ORR), disease control rate (DCR), and overall survival (OS) of these patients? What is the safety and tolerability profile of this combined treatment? Which molecular biomarkers can predict the efficacy of this therapy? Eligible subjects (who have signed informed consent) will receive RALOX hepatic artery infusion chemotherapy plus QL1706 (7.5mg, intravenous infusion every 3 weeks) and bevacizumab (15mg/kg, intravenous infusion every 3 weeks), with 3 weeks as one treatment cycle. Treatment will continue until a protocol-specified discontinuation event occurs. After treatment, subjects will undergo post-treatment safety follow-up and survival follow-up; those who discontinue treatment for reasons other than disease progression or death will also have tumor progression follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form;
2. Aged ≥ 18 years, male and female subjects are both eligible;
3. Clinically or pathologically confirmed hepatocellular carcinoma (HCC), with no prior systemic anti-tumor therapy for HCC (including but not limited to molecular targeted therapy, systemic chemotherapy, immunotherapy such as anti-PD-1/PD-L1/CTLA-4 monoclonal antibodies, etc.);
4. Complicated with Type VP3 or VP4 portal vein tumor thrombosis (PVTT);
5. Confirmed to have at least one measurable target lesion by imaging examination during the screening period in accordance with RECIST v1.1 criteria. The measurable lesions should not have received local treatment such as radiotherapy (lesions within the area of previous local treatment can also be selected as target lesions if disease progression is confirmed);
6. Child-Pugh score ≤ 7 points (Child-Pugh class A-B);
7. The maximum diameter of liver tumor ≥ 7 cm;
8. ECOG performance status 0 to 1;
9. Expected survival time ≥ 12 weeks;
10. Function of vital organs meeting the following requirements:

Absolute neutrophil count (ANC) ≥ 1.5×10⁹/L; Platelet count ≥ 50×10⁹/L; Hemoglobin ≥ 90 g/L; Serum albumin ≥ 29 g/L; Bilirubin ≤ 2 × upper limit of normal (ULN); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 5 × ULN, alkaline phosphatase (AKP) ≤ 5 × ULN; Serum creatinine ≤ 1.5 × ULN or creatinine clearance rate (CrCl) ≥ 50 mL/min calculated by the Cockcroft-Gault formula; 11.Eligible patients with reproductive potential (males and females) must agree to use a reliable contraceptive method (hormonal, barrier method or abstinence) with their partners during the trial and for at least 180 days after the last dose; female patients of childbearing potential must have a negative serum pregnancy test within 7 days prior to the first study medication administration.

Exclusion Criteria:

1. Histologically or cytologically confirmed fibrolamellar hepatocellular carcinoma, sarcomatoid hepatocellular carcinoma, cholangiocellular carcinoma, mixed hepatocellular carcinoma, etc.;
2. Active autoimmune disease, or a history of autoimmune disease with potential for recurrence (including but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism [patients whose condition is controllable only with hormone replacement therapy are not excluded]); Note: Patients with dermatological diseases that do not require systemic treatment (e.g., vitiligo, psoriasis, alopecia), type 1 diabetes with good glycemic control under insulin therapy, or asthma that achieved complete remission in childhood and requires no intervention in adulthood are eligible for enrollment; patients with asthma requiring medical intervention with bronchodilators are ineligible.
3. Administration of immunosuppressants or systemic hormonal therapy for immunosuppressive purposes within 2 weeks prior to the first study medication (dose > 10 mg/day prednisone or an equivalent dose of other hormones);
4. Current interstitial pneumonia or interstitial lung disease, a history of interstitial pneumonia or interstitial lung disease requiring hormonal therapy, or other pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), pneumoconiosis, drug-related pneumonia, idiopathic pneumonia that may interfere with the judgment and management of immune-related pulmonary toxicity; patients with evidence of active pneumonia on screening CT or severe impairment of pulmonary function are excluded. Radiation pneumonitis within the radiation field is permitted;
5. Confirmed active pulmonary tuberculosis. For subjects with suspected active pulmonary tuberculosis, a definitive diagnosis shall be made based on chest imaging, sputum examination, and clinical symptoms and signs;
6. Known hypersensitivity to the active ingredients or excipients of the study drugs, or a history of severe hypersensitivity to any other monoclonal antibody or anti-angiogenic targeted drugs;
7. Known history of central nervous system (CNS) metastasis or hepatic encephalopathy;
8. A history of allogeneic stem cell transplantation or solid organ transplantation;
9. Moderate to severe ascites with clinical symptoms requiring therapeutic paracentesis or drainage (except for patients with only a small amount of ascites shown by imaging without clinical symptoms), or uncontrolled moderate to large pleural effusion or pericardial effusion;
10. Severe cardiovascular and cerebrovascular diseases, including but not limited to:

(1) Severe cardiac rhythm or conduction abnormalities (e.g., ventricular or supraventricular arrhythmias requiring clinical intervention, grade Ⅱ-Ⅲ atrioventricular block), QTcF interval ≥ 450 ms (males) or QTcF interval ≥ 470 ms (females) (if the QTcF interval is abnormal at screening, two additional tests shall be performed at an interval of at least 5 minutes, and the average value shall be taken); unstable angina pectoris, etc.; (2) Acute coronary syndrome, congestive heart failure, aortic dissection, stroke, transient ischemic attack (TIA) or other grade 3 and above cardiovascular and cerebrovascular events within 6 months prior to the first study medication; (3) New York Heart Association (NYHA) cardiac function classification ≥ grade II or left ventricular ejection fraction (LVEF) < 50%; (4) Poorly controlled hypertension (systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg after treatment with two or more antihypertensive drugs); 11.Coagulation dysfunction (INR > 2.0, prothrombin time (PT) prolonged by more than 6 seconds), with obvious bleeding tendency or other evidence of major coagulation disorders: clinically significant hemoptysis or tumor bleeding of any cause within 2 weeks prior to the first study medication; a history of thrombosis or embolism within 6 months prior to the first study medication; therapeutic anticoagulant therapy (except low-molecular-weight heparin) within 2 weeks prior to the first study medication; or antiplatelet therapy (e.g., aspirin > 325 mg/day, clopidogrel > 75 mg/day, dipyridamole, ticlopidine, cilostazol) within 10 days prior to the first study medication, or patients requiring long-term antiplatelet therapy; patients with metastatic lesions invading large blood vessels, respiratory tract or middle mediastinum with a significant risk of bleeding; 12.A history of esophageal or gastric variceal bleeding caused by portal hypertension within 6 months prior to the first study medication; confirmed severe varices by endoscopy within 3 months prior to the first study medication; or evidence of portal hypertension (including splenomegaly detected by imaging) with a high risk of bleeding assessed by the investigator (including moderate to severe esophagogastric varices with bleeding risk, active local peptic ulcer, and persistent positive fecal occult blood, which require gastroscopy to exclude patients with "red signs". Patients with a history of "red signs" on gastroscopy are excluded); 13.Any life-threatening bleeding event within 3 months prior to the first study medication, including those requiring blood transfusion, surgery or local treatment, and continuous drug therapy; 14.A history of abdominal fistula, gastrointestinal perforation or abdominal abscess within 6 months prior to the first study medication; 15.A history of intestinal obstruction and/or clinical signs or symptoms of gastrointestinal obstruction within 6 months prior to the first study medication, including incomplete obstruction related to the primary disease or requiring routine parenteral hydration, parenteral nutrition or tube feeding; 16.Severe unhealed wounds, active ulcers or untreated fractures; 17.Urinalysis showing urine protein ≥ ++ with a confirmed 24-hour urine protein excretion > 1.0 g; 18.Severe infection within 4 weeks prior to the first study medication (including but not limited to hospitalization due to infection, bacteremia or severe pneumonia complications); active infection requiring oral or intravenous therapeutic antibiotics within 2 weeks prior to the first study medication (patients receiving prophylactic antibiotics, e.g., for prevention of urinary tract infection or acute exacerbation of chronic obstructive pulmonary disease, are eligible); unexplained fever ≥ 38.5℃ within 7 days prior to medication administration, or baseline white blood cell count > 15×10⁹/L; 19.Congenital or acquired immune deficiency (e.g., HIV-infected patients), or confirmed active syphilis infection; 20.A history of other malignant tumors except HCC within 5 years prior to the first study medication or concurrent malignant tumors. Patients with the following cured localized tumors are eligible for enrollment: basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, carcinoma in situ of the prostate, carcinoma in situ of the cervix, carcinoma in situ of the breast, etc.; 21.Hepatic surgery, local treatment for HCC or investigational drug therapy within 4 weeks prior to the first study medication; administration of traditional Chinese medicine preparations with anti-HCC effects within 2 weeks prior to the first study medication; or toxic reactions caused by previous treatment (except alopecia) that have not recovered to ≤ grade 1 (per NCI-CTCAE v5.0); 22.Administration of drugs with immunomodulatory effects (including but not limited to interferon, interleukin) within 2 weeks prior to the first study medication; 23.Participation in other clinical studies and administration of other investigational drugs within 4 weeks prior to the first study medication; 24.Administration of live attenuated vaccines within 4 weeks prior to the first study medication, or anticipated need for such vaccination during the study treatment or within 90 days after the last study medication; 25.Major surgery (except for diagnostic purposes) within 4 weeks prior to the first study medication, or anticipated major surgery during the study period (major surgery is defined as surgery performed under general anesthesia that requires a recovery period of at least 3 weeks before initiation of study drug treatment); tissue biopsy or other minor surgical procedures within 7 days prior to the first study medication, except for venous catheterization for intravenous infusion; 26.Pregnant or lactating women, or women of childbearing potential who refuse to take contraceptive measures; 27.Other factors judged by the investigator that may affect the study results or lead to forced early termination of the study, such as alcoholism, drug abuse, other severe diseases (including mental illness) requiring combined treatment, severe abnormal laboratory tests, or family/social factors that may affect patient safety.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-12-25 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival time (PFS) | From date of first dose of study drug to the date of first documentation of disease progression or death, whichever occurs first (up to approximately 2 years)
  The progression free survival time defined as the time from the first study dose date to the date of first documentation of disease progression as assessed by RECIST 1.1

SECONDARY OUTCOMES:
Objective response rate (ORR) | From date of first dose of study drug until disease progression, development of unacceptable toxicity, withdrawal of consent, or sponsor termination (up to approximately 2 years)
The disease control rate (DCR) | From date of first dose of study drug until disease progression, stable disease, development of unacceptable toxicity, withdrawal of consent, or sponsor termination (up to approximately 2 years)
Overall survival time (OS) | From date of first dose of study drug to the date of first documentation of disease progression or death, whichever occurs first (up to approximately 2 years)
Treatment-Emergent Adverse Events (Safety and Tolerability) | Throughout the entire treatment period and 30 days after the last dose

CONTACTS AND LOCATIONS:
Overall Officials: Jinzhang Chen, Study Director, Study Director — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong, China